CLINICAL TRIAL: NCT04545606
Title: Targeting Insomnia in School Aged Children With Autism Spectrum Disorder
Acronym: RECHArge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christina McCrae, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019182; W81XW-H2010399 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-08-26; First posted 2020-09-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Insomnia Chronic; Autism Spectrum Disorder
Keywords: cognitive behavioral therapy, behavioral therapy; children
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person CBT for insomnia in children with autism (Experimental): In-person cognitive-behavioral treatment (CBT) for insomnia in children with autism will be conducted at the Thompson Center. In-person treatment will consist of four 50-minute, individually administered sessions and four bi-monthly, 20-minute telephone boosters. Using a flexible, case conceptualization approach, the therapist will adapt the treatment to parent and child characteristics (i.e., verbal skills, development) and family situation/dynamics - promoting optimal efficacy and enhancing broad clinical applicability. Module administration order will be tailored to prioritize each child/family's most pressing sleep concerns based on the clinical interview.
  Interventions: Behavioral: In-Person CBT for insomnia in children with autism
- Remote CBT for insomnia in children with autism (Experimental): Remote/videoconferenced cognitive-behavioral treatment (CBT) for insomnia in children with autism will be conducted from home (families)/Thompson Center (therapist). Remote treatment will consist of four 50-minute, individually administered sessions and four bi-monthly, 20-minute telephone boosters. Using a flexible, case conceptualization approach, the therapist will adapt the treatment to parent and child characteristics (i.e., verbal skills, development) and family situation/dynamics - promoting optimal efficacy and enhancing broad clinical applicability. Module administration order will be tailored to prioritize each child/family's most pressing sleep concerns based on the clinical interview.
  Interventions: Behavioral: Remote CBT for insomnia in children with autism
- Remote behavioral SHARE for insomnia in children with autism (Experimental): Remote/videoconferenced behavioral sleep hygiene and related education (SHARE) for insomnia in children with autism will be conducted from home (families)/Thompson Center (therapist). Remote treatment will consist of four 50-minute, individually administered sessions and four bi-monthly, 20-minute telephone boosters. Using a flexible, case conceptualization approach, the therapist will adapt the treatment to parent and child characteristics (i.e., verbal skills, development) and family situation/dynamics - promoting optimal efficacy and enhancing broad clinical applicability. Module administration order will be tailored to prioritize each child/family's most pressing sleep and related health related concerns/interests.
  Interventions: Behavioral: Remote sleep hygiene and related education (SHARE) for insomnia in children with autism

INTERVENTIONS:
Behavioral: In-Person CBT for insomnia in children with autism — 7 modules administered in-person
  1. Sleep Hygiene & Sleep Prescription
  2. Bedtime Routine & Parent Management
  3. Cue Control & Parent Management
  4. Co-Sleeping & Parents Fading out of Room
  5. Circadian Education, Morning Routine, & Relaxation
  6. Cognitive Therapy Basics
  7. Nighttime Fears, Anxiety, & Nightmares
  Arms: In-person CBT for insomnia in children with autism
Behavioral: Remote CBT for insomnia in children with autism — 7 modules administered over telehealth/videoconferencing
  1. Sleep Hygiene & Sleep Prescription
  2. Bedtime Routine & Parent Management
  3. Cue Control & Parent Management
  4. Co-Sleeping & Parents Fading out of Room
  5. Circadian Education, Morning Routine, & Relaxation
  6. Cognitive Therapy Basics
  7. Nighttime Fears, Anxiety, & Nightmares
  Arms: Remote CBT for insomnia in children with autism
Behavioral: Remote sleep hygiene and related education (SHARE) for insomnia in children with autism — 7 modules administered over telehealth/videoconferencing
  1. Sleep Education
  2. Sleep Architecture & Parasomnias
  3. Physical Activity & Sleep
  4. Nutrition, My Plate, & Breathing during Sleep
  5. Stress, Sleep, Dreams, & Nightmares Connections
  6. Mood, Self-Esteem, & Sleep
  7. Light & Dark Cycle
  Arms: Remote behavioral SHARE for insomnia in children with autism

SUMMARY:
Children with Autism Spectrum Disorder (ASD) and insomnia, and their parent(s) will undergo 4 sessions of behavioral therapy for sleep problems followed by 4 bimonthly booster sessions. Children and their families will be randomly assigned to one of three conditions: cognitive behavioral therapy (in-person), cognitive behavioral therapy (remote), or behavioral therapy (remote). Arousal will be measured through heart-rate variability. Sleep and secondary outcomes (child daytime behavior, parent sleep) will be collected at baseline (weeks 1-2 before starting the treatment), post-treatment (weeks 6-8 from baseline), 6-month follow-up, and 12-month follow-up.

DETAILED DESCRIPTION:
Children with autism often have difficulties falling and staying asleep at night. Those sleep difficulties can contribute to daytime problems with irritability, learning, and behavior. Parents are often stressed about their child's sleep difficulties and as a result, their sleep can suffer as well. Treatment that focuses on establishing behaviors and routines that help reduce arousal and support good sleep are helpful for improving the sleep of children without autism, but have not yet been tested in children with autism.

Previous studies have indicated that distance can make it difficult for families to participate in treatment. As such, we will conduct treatment remotely for two of treatment arms. Having remote versions of the treatment can expand the number of children and families that are able to receive these promising treatments. This may be particularly important for children with ASD living in rural and underserved areas as well as those in military families that may not have access to a healthcare provider with training in behavioral sleep treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1) 6-12a yrs
* 2) Verbal IQ >= 70
* 3) participation of child's parent or legal guardian living in the same home
* 4) parent/guardian ability to read and understand English at the 5th-grade level
* 5) child diagnosed with ASD and insomnia

ASD:

* 1) previous DSM diagnosis of ASD
* 2) evaluation using gold-standard diagnostic tools (i.e., Autism Diagnostic Observation Schedule (ADOS) and/or Autism Diagnostic Interview-Revised [ADI-R])

Insomnia:

* 1) complaints of difficulties falling asleep, staying asleep, or early morning awakening by child report or parent observation for 3+ mos
* 2) daytime dysfunction (mood, cognitive, social, academic) due to insomnia
* 3) baseline diaries and actigraphy indicate >30 mins. of sleep onset latency, wake after sleep onset, or early morning awakening (time between last awakening and out of bed time) on 6+ nights

Exclusion Criteria:

* 1) parent unable to provide informed consent or child unable to provide assent
* 2) unwilling to accept random assignment
* 3) participation in another randomized research project
* 4) parent unable to complete forms or implement treatment procedures due to cognitive impairment
* 5) untreated medical comorbidity, including other sleep disorders (e.g., apnea, epilepsy, psychotic disorders, suicidal ideation/intent, [frequent] parasomnias)
* 6) psychotropic or other medications that alter sleep with the exceptions of stimulants, sleep medications, and/or melatonin as described in #7 (see Notes below for details)
* 7) stimulants, sleep medications (prescribed or OTC), and/or melatonin within the last 1 month (unless stabilized on medication for 3+ months)
* 8) participation in non-pharmacological treatment (including CBT) for sleep outside current trial
* 9) parent report of inability to undergo Holter Monitoring or actigraphy (e.g., extreme sensitivity, behavioral outbursts)
* 10) other conditions adversely affecting trial participation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Baseline Average Objective Sleep Efficiency for the child | 24/7 during each 2 week assessment at Baseline
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Sleep Efficiency for the child from baseline to immediately after the intervention | 24/7 during each 2 week assessment immediately after the intervention
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Sleep Efficiency for the child from baseline to 6 months | 24/7 during each 2 week assessment at 6 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Sleep Efficiency for the child from baseline to 12 months | 24/7 during each 2 week assessment at 12 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Baseline Average Bed/Waketime Variability for the child | 24/7 during each 2 week assessment at Baseline
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity and daily diary report
Change in Average Bed/Waketime Variability for the child from baseline to immediately after the intervention | 24/7 during each 2 week assessment immediately after the intervention
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity and daily diary report
Change in Average Bed/Waketime Variability for the child from baseline to 6 months | 24/7 during each 2 week assessment at 6 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity and daily diary report
Change in Average Bed/Waketime Variability for the child from baseline to 12 months | 24/7 during each 2 week assessment at 12 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity and daily diary report
Baseline Average RMSDNN (root mean squared st. dev. of N-N intervals) for the child | 8 minute protocol during rest at Baseline (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the child from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the child from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the child from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Baseline Average Objective Total Sleep Time for the parent | 24/7 during each 2 week assessment at Baseline
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Total Sleep Time for the parent from baseline to immediately after the intervention | 24/7 during each 2 week assessment immediately after the intervention
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Total Sleep Time for the parent from baseline to 6 months | 24/7 during each 2 week assessment at 6 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity
Change in Average Objective Total Sleep Time for the parent from baseline to 12 months | 24/7 during each 2 week assessment at 12 month follow up
  Actigraph (Actiwatch 2â, Philips Respironics) measures light and gross motor activity

SECONDARY OUTCOMES:
Baseline Aberrant Behavior Checklist (ABC) for the child | Baseline
  Aberrant Behavior Checklist (ABC) is a 58-item parent-report measure of daytime problem behaviors that is psychometrically strong and sensitive to treatment effects in children with ASD. It will be filled out by the parent in reference to the child.
Aberrant Behavior Checklist (ABC) for the child immediately after the intervention | Immediately after the intervention
  Aberrant Behavior Checklist (ABC) is a 58-item parent-report measure of daytime problem behaviors that is psychometrically strong and sensitive to treatment effects in children with ASD. It will be filled out by the parent in reference to the child.
Aberrant Behavior Checklist (ABC) for the child at 6 months | At 6 month follow up
  Aberrant Behavior Checklist (ABC) is a 58-item parent-report measure of daytime problem behaviors that is psychometrically strong and sensitive to treatment effects in children with ASD. It will be filled out by the parent in reference to the child.
Aberrant Behavior Checklist (ABC) for the child at 12 months | At 12 month follow up
  Aberrant Behavior Checklist (ABC) is a 58-item parent-report measure of daytime problem behaviors that is psychometrically strong and sensitive to treatment effects in children with ASD. It will be filled out by the parent in reference to the child.
Baseline Conners' Continuous Performance Test - 3rd Edition (CCPT-3) for a child (ages 8+) | Baseline
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Continuous Performance Test - 3rd Edition (CCPT-3) for a child (ages 8+) immediately after the intervention | Immediately after the intervention
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Continuous Performance Test - 3rd Edition (CCPT-3) for a child (ages 8+) at 6 months | At 6 month follow up
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Continuous Performance Test - 3rd Edition (CCPT-3) for a child (ages 8+) at 12 months | At 12 month follow up
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Baseline Conners' Kiddie Continuous Performance Test (K-CPT) for a child (ages 6-7) | Baseline
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Kiddie Continuous Performance Test (K-CPT) for a child (ages 6-7) immediately after the intervention | Immediately after the intervention
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Kiddie Continuous Performance Test (K-CPT) for a child (ages 6-7) at 6 months | At 6 month follow up
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Conners' Kiddie Continuous Performance Test (K-CPT) for a child (ages 6-7) at 12 months | At 12 month follow up
  Conners' Continuous Performance Test - 3rd Edition (CCPT-3) is a computerized measure of inattentiveness, impulsivity, sustained attention, and vigilance for aged 8 and above. Conners' Kiddie Continuous Performance Test (K-CPT) will be used for children aged 6 and 7 which provides a comparable measure of the four domains of attention. To account for two different measures in analyses, standardized scores will be used.
Baseline Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) for the child | Baseline
  Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) is a 86-item parent-report measure of day-to-day executive functioning and impairment. It will be filled out by the parent in reference to the child.
Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) for the child immediately after the intervention | Immediately after the intervention
  Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) is a 86-item parent-report measure of day-to-day executive functioning and impairment. It will be filled out by the parent in reference to the child.
Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) for the child at 6 months | At 6 month follow up
  Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) is a 86-item parent-report measure of day-to-day executive functioning and impairment. It will be filled out by the parent in reference to the child.
Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) for the child at 12 months | At 12 month follow up
  Behavior Rating Inventory of Executive Function - 2nd Edition (BRIEF-2) is a 86-item parent-report measure of day-to-day executive functioning and impairment. It will be filled out by the parent in reference to the child.
Baseline Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) for the child | Baseline
  Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) includes 20 parent-reported items and is an appropriate outcome tool for children with ASD. It will be filled out by the parent in reference to the child.
Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) for the child immediately after the intervention | Immediately after the intervention
  Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) includes 20 parent-reported items and is an appropriate outcome tool for children with ASD. It will be filled out by the parent in reference to the child.
Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) for the child at 6 months | At 6 month follow up
  Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) includes 20 parent-reported items and is an appropriate outcome tool for children with ASD. It will be filled out by the parent in reference to the child.
Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) for the child at 12 months | At 12 month follow up
  Child and Adolescent Symptom Inventory - 4th Edition Revised (CASI-4R) includes 20 parent-reported items and is an appropriate outcome tool for children with ASD. It will be filled out by the parent in reference to the child.
Baseline Child Quality of Life: PedsQL Child Form for the child | Baseline
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the child in reference to the child.
Child Quality of Life: PedsQL Child Form for the child immediately after the intervention | Immediately after the intervention
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the child in reference to the child.
Child Quality of Life: PedsQL Child Form for the child at 6 months | At 6 month follow up
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the child in reference to the child.
Child Quality of Life: PedsQL Child Form for the child at 12 months | At 12 month follow up
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the child in reference to the child.
Baseline Child Quality of Life: PedsQL Parent Form for the child | Baseline
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the parent in reference to the child.
Child Quality of Life: PedsQL Parent Form for the child immediately after the intervention | Immediately after the intervention
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the parent in reference to the child.
Child Quality of Life: PedsQL Parent Form for the child at 6 months | At 6 month follow up
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the parent in reference to the child.
Child Quality of Life: PedsQL Parent Form for the child at 12 months | At 12 month follow up
  Child Quality of Life: PedsQL is a 23-item scale measuring children's QOL. It has excellent internal consistency, clinical validity, and factor-analytic support. It will be filled out by the parent in reference to the child.
Baseline Average Subjective Sleep Onset Latency for the child | Each morning for 2 weeks at Baseline
  Diary-reported amount of time from lights out to beginning of sleep filled out by the child (with parent help) regarding the child's sleep
Change in Average Subjective Sleep Onset Latency for the child from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported amount of time from lights out to beginning of sleep filled out by the child (with parent help) regarding the child's sleep
Change in Average Subjective Sleep Onset Latency for the child from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported amount of time from lights out to beginning of sleep filled out by the child (with parent help) regarding the child's sleep
Change in Average Subjective Sleep Onset Latency for the child from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported amount of time from lights out to beginning of sleep filled out by the child (with parent help) regarding the child's sleep
Baseline Average Subjective Total Wake Time for the child | Each morning for 2 weeks at Baseline
  Diary-reported time awake from lights out until out of bed filled out by the child (with a parent's help) regarding the child's sleep
Change in Average Subjective Total Wake Time for the child from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported time awake from lights out until out of bed filled out by the child (with a parent's help) regarding the child's sleep
Change in Average Subjective Total Wake Time for the child from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported time awake from lights out until out of bed filled out by the child (with a parent's help) regarding the child's sleep
Change in Average Subjective Total Wake Time for the child from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported time awake from lights out until out of bed filled out by the child (with a parent's help) regarding the child's sleep
Baseline Average Subjective Total Sleep Time for the child | Each morning for 2 weeks at Baseline
  Diary-reported total sleep time filled out by the child (with help of a parent) regarding the child's sleep
Change in Average Subjective Total Sleep Time for the child from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported total sleep time filled out by the child (with help of a parent) regarding the child's sleep
Change in Average Subjective Total Sleep Time for the child from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported total sleep time filled out by the child (with help of a parent) regarding the child's sleep
Change in Average Subjective Total Sleep Time for the child from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported total sleep time filled out by the child (with help of a parent) regarding the child's sleep
Baseline Average Subjective Sleep Efficiency for the child | Each morning for 2 weeks at Baseline
  Diary-reported total sleep time/time in bed x 100% filled out by the child (with help from a parent) regarding the child's sleep
Change in Average Subjective Sleep Efficiency for the child from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported total sleep time/time in bed x 100% filled out by the child (with help from a parent) regarding the child's sleep
Change in Average Subjective Sleep Efficiency for the child from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported total sleep time/time in bed x 100% filled out by the child (with help from a parent) regarding the child's sleep
Change in Average Subjective Sleep Efficiency for the child from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported total sleep time/time in bed x 100% filled out by the child (with help from a parent) regarding the child's sleep
Baseline Average LF/HF ratio for the child | 8 minute protocol during rest at Baseline (in clinic)
  An index of the child's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the child from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  An index of the child's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the child from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  An index of the child's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the child from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  An index of the child's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Baseline Average pNN50 (% of N-N intervals > 50 ms) for the child | 8 minute protocol during rest at Baseline (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the child from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the child from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the child from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  Child arousal measured by Holter Monitors, 8 min ECG
Baseline Average LF/HF ratio for the parent | 8 minute protocol during rest at Baseline (in clinic)
  An index of the parent's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the parent from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  An index of the parent's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the parent from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  An index of the parent's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Change in Average LF/HF ratio for the parent from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  An index of the parent's autonomic nervous system regulation measured by Holter Monitors, 8 min ECG
Baseline Average pNN50 (% of N-N intervals > 50 ms) for the parent | 8 minute protocol during rest at Baseline (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the parent from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the parent from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average pNN50 (% of N-N intervals > 50 ms) for the parent from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Baseline Average RMSDNN (root mean squared st. dev. of N-N intervals) for the parent | 8 minute protocol during rest at Baseline (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the parent from baseline to immediately after the intervention | 8 minute protocol during rest immediately after the intervention (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the parent from baseline to 6 months | 8 minute protocol during rest at 6 month follow up (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Change in Average RMSDNN (root mean squared st. dev. of N-N intervals) for the parent from baseline to 12 months | 8 minute protocol during rest at 12 month follow up (in clinic)
  Parent arousal measured by Holter Monitors, 8 min ECG
Baseline State-Trait Anxiety Inventory (STAI-Y1) for the parent | Baseline
  State-Trait Anxiety Inventory (STAI-Y1) includes 20 self-descriptive statements rated according to how the parent generally feels on a 4-point scale [1 (not at all) to 4 (very much so)]. This will be filled out by the parents regarding the parents.
State-Trait Anxiety Inventory (STAI-Y1) for the parent immediately after the intervention | Immediately after the intervention
  State-Trait Anxiety Inventory (STAI-Y1) includes 20 self-descriptive statements rated according to how the parent generally feels on a 4-point scale [1 (not at all) to 4 (very much so)]. This will be filled out by the parents regarding the parents.
State-Trait Anxiety Inventory (STAI-Y1) for the parent at 6 months | At 6 month follow up
  State-Trait Anxiety Inventory (STAI-Y1) includes 20 self-descriptive statements rated according to how the parent generally feels on a 4-point scale [1 (not at all) to 4 (very much so)]. This will be filled out by the parents regarding the parents.
State-Trait Anxiety Inventory (STAI-Y1) for the parent at 12 months | At 12 month follow up
  State-Trait Anxiety Inventory (STAI-Y1) includes 20 self-descriptive statements rated according to how the parent generally feels on a 4-point scale [1 (not at all) to 4 (very much so)]. This will be filled out by the parents regarding the parents.
Baseline Beck Depression Inventory (BDI-II) for the parent | Baseline
  Beck Depression Inventory (BDI-II) includes 21 items that measures the severity of depressive symptomatology on a 4-point scale (0-absence of symptoms; 3-severe). This will be filled out by the parents regarding the parents.
Beck Depression Inventory (BDI-II) for the parent immediately after the intervention | Immediately after the intervention
  Beck Depression Inventory (BDI-II) includes 21 items that measures the severity of depressive symptomatology on a 4-point scale (0-absence of symptoms; 3-severe). This will be filled out by the parents regarding the parents.
Beck Depression Inventory (BDI-II) for the parent at 6 months | At 6 month follow up
  Beck Depression Inventory (BDI-II) includes 21 items that measures the severity of depressive symptomatology on a 4-point scale (0-absence of symptoms; 3-severe). This will be filled out by the parents regarding the parents.
Beck Depression Inventory (BDI-II) for the parent at 12 months | At 12 month follow up
  Beck Depression Inventory (BDI-II) includes 21 items that measures the severity of depressive symptomatology on a 4-point scale (0-absence of symptoms; 3-severe). This will be filled out by the parents regarding the parents.
Baseline Fatigue Severity Scale for the parent | Baseline
  Fatigue Severity Scale includes 9 items on the severity of fatigue and how fatigue interferes with activities on a 7-point scale (1-strongly disagree; 7-strongly agree). This will be filled out by the parents regarding the parents.
Fatigue Severity Scale for the parent immediately after the intervention | Immediately after the intervention
  Fatigue Severity Scale includes 9 items on the severity of fatigue and how fatigue interferes with activities on a 7-point scale (1-strongly disagree; 7-strongly agree). This will be filled out by the parents regarding the parents.
Fatigue Severity Scale for the parent at 6 months | At 6 month follow up
  Fatigue Severity Scale includes 9 items on the severity of fatigue and how fatigue interferes with activities on a 7-point scale (1-strongly disagree; 7-strongly agree). This will be filled out by the parents regarding the parents.
Fatigue Severity Scale for the parent at 12 months | At 12 month follow up
  Fatigue Severity Scale includes 9 items on the severity of fatigue and how fatigue interferes with activities on a 7-point scale (1-strongly disagree; 7-strongly agree). This will be filled out by the parents regarding the parents.
Baseline Daily Fatigue for the parent | Baseline
  Daily Fatigue rated on electronic diaries (0-none;100-most intense imaginable). This will be filled out by the parents regarding the parents.
Daily Fatigue for the parent immediately after the intervention | Immediately after the intervention
  Daily Fatigue rated on electronic diaries (0-none;100-most intense imaginable). This will be filled out by the parents regarding the parents.
Daily Fatigue for the parent at 6 months | At 6 month follow up
  Daily Fatigue rated on electronic diaries (0-none;100-most intense imaginable). This will be filled out by the parents regarding the parents.
Daily Fatigue for the parent at 12 months | At 12 month follow up
  Daily Fatigue rated on electronic diaries (0-none;100-most intense imaginable). This will be filled out by the parents regarding the parents.
Baseline Caregiver Strain Index (CSI) for the parent | Baseline
  Caregiver Strain Index (CSI) includes 12 items on caregiving impact on well-being. This will be filled out by the parents regarding the parents.
Caregiver Strain Index (CSI) for the parent immediately after the intervention | Immediately after the intervention
  Caregiver Strain Index (CSI) includes 12 items on caregiving impact on well-being. This will be filled out by the parents regarding the parents.
Caregiver Strain Index (CSI) for the parent at 6 months | At 6 month follow up
  Caregiver Strain Index (CSI) includes 12 items on caregiving impact on well-being. This will be filled out by the parents regarding the parents.
Caregiver Strain Index (CSI) for the parent at 12 months | At 12 month follow up
  Caregiver Strain Index (CSI) includes 12 items on caregiving impact on well-being. This will be filled out by the parents regarding the parents.
Baseline Average Subjective Sleep Onset Latency for the parent | Each morning for 2 weeks at Baseline
  Diary-reported amount of time from lights out to beginning of sleep filled out by the parent regarding parent sleep
Change in Average Subjective Sleep Onset Latency for the parent from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported amount of time from lights out to beginning of sleep filled out by the parent regarding parent sleep
Change in Average Subjective Sleep Onset Latency for the parent from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported amount of time from lights out to beginning of sleep filled out by the parent regarding parent sleep
Change in Average Subjective Sleep Onset Latency for the parent from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported amount of time from lights out to beginning of sleep filled out by the parent regarding parent sleep
Baseline Average Subjective Total Wake Time for the parent | Each morning for 2 weeks at Baseline
  Diary-reported time awake from lights out until out of bed filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Wake Time for the parent from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported time awake from lights out until out of bed filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Wake Time for the parent from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported time awake from lights out until out of bed filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Wake Time for the parent from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported time awake from lights out until out of bed filled out by the parent regarding the parent's sleep
Baseline Average Subjective Total Sleep Time for the parent | Each morning for 2 weeks at Baseline
  Diary-reported total sleep time filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Sleep Time for the parent from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported total sleep time filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Sleep Time for the parent from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported total sleep time filled out by the parent regarding the parent's sleep
Change in Average Subjective Total Sleep Time for the parent from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported total sleep time filled out by the parent regarding the parent's sleep
Baseline Average Subjective Sleep Efficiency for the parent | Each morning for 2 weeks at Baseline
  Diary-reported total sleep time/time in bed x 100% filled out by the parent regarding the parent's sleep
Change in Average Subjective Sleep Efficiency for the parent from baseline to immediately after the intervention | Each morning for 2 weeks immediately after the intervention
  Diary-reported total sleep time/time in bed x 100% filled out by the parent regarding the parent's sleep
Change in Average Subjective Sleep Efficiency for the parent from baseline to 6 months | Each morning for 2 weeks at 6 month follow up
  Diary-reported total sleep time/time in bed x 100% filled out by the parent regarding the parent's sleep
Change in Average Subjective Sleep Efficiency for the parent from baseline to 12 months | Each morning for 2 weeks at 12 month follow up
  Diary-reported total sleep time/time in bed x 100% filled out by the parent regarding the parent's sleep

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Thompson Center for Autism and Neurodevelopmental Disorders, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the research team to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared after data collection is complete and results have been published.
Access Criteria: De-identified data will be made available to other qualified investigators who aim to verify data, conduct meta-analyses, or collaborate with the research team on analyses that are not already planned.

REFERENCES:
- [Derived] McCrae CS, Mazurek MO, Curtis AF, Beversdorf DQ, Deroche CB, Golzy M, Sohl KA, Ner ZH, Davis BE, Stearns MA, Nair N. Protocol for targeting insomnia in school-aged children with autism spectrum disorder without intellectual disability: a randomised control trial. BMJ Open. 2021 Aug 25;11(8):e045944. doi: 10.1136/bmjopen-2020-045944. PMID 34433593